CLINICAL TRIAL: NCT01906255
Title: Adherence, HIV-1 Infection, Resistance, and Renal and Skeletal Adverse Event in Individuals Taking Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF, Truvada®) for HIV Pre-Exposure Prophylaxis (PrEP): A Pooled Observational Study
Brief Title: Adherence, HIV-1 Infection, Resistance, and Renal and Skeletal Adverse Event in Individuals Taking Truvada® for HIV Pre-Exposure Prophylaxis (PrEP)
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-276-0104; EUPAS24332 (Registry Identifier: ENCePP)
Record Dates: First submitted 2013-07-15; First posted 2013-07-24 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: HIV
Keywords: HIV-1; Truvada; FTC/TDF; Pre-exposure prophylaxis; PrEP; Adherence; Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FTC/TDF for PrEP: HIV-1 negative adults (any sex/gender, including transgender, pregnancy) who are participating in observational or clinical studies on FTC/TDF for PrEP

SUMMARY:
This is an observational study of HIV-1 negative individuals who participated in demonstration projects or clinical studies and took daily Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF, Truvada®) for pre-exposure prophylaxis (PrEP). All individuals were enrolled and followed as described in the parent PrEP demonstration project or clinical study protocol until study completion, HIV-1 infection, discontinuation due to an adverse event, lost to follow-up, or administrative censoring.

In the protocols of the parent PrEP observational or clinical studies, participants had follow-up visits on average every 3 months for evaluation of adherence, renal and bone adverse events, and HIV-1 infection status. Adherence was determined by the specific FTC/TDF drug level measurement(s) outlined in the parent protocol.

Gilead had collected data from 21 global PrEP demonstration projects and clinical studies for over 7,000 Truvada for PrEP users who had at least one measurement of adherence. Data from the different contributing studies were pooled for statistical analyses by Gilead.

ELIGIBILITY:
Inclusion Criteria:

* Participants in an FTC/TDF for PrEP observational or clinical study
* HIV-1 negative individual at the time of enrollment in a demonstration project or clinical study
* Participants with at least one measurement of tenofovir-diphosphate (TFV-DP) in dried blood spot (DBS) or tenofovir (TFV) in plasma

Exclusion Criteria:

* This is an observational study and will collect HIV-1 infection and resistance information along with renal or skeletal adverse events without intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seven thousand (7000) HIV-1 negative adults (any sex/gender, including transgender, pregnancy) who are participating in observational or clinical studies on FTC/TDF for PrEP
Sampling Method: Non-Probability Sample
Enrollment: 10577 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Treatment adherence, as measured by drug level, to the once-daily dosing regimen of FTC/TDF for PrEP | Baseline to Year 3

SECONDARY OUTCOMES:
Time to onset of signs and/or symptoms of acute HIV infection before and after seroconversion during treatment | Baseline to Year 3
  The time to onset of signs and/or symptoms if acute HIV infection in relation to exposure to study drug will be recorded. Signs and symptoms include fever, lymphadenopathy, pharyngitis, rash, myalgia, malaise, mouth and esophageal sores, and may also include, but less commonly, headache, nausea and vomiting, enlarged liver/spleen, weight loss, thrush, and neurological symptoms.
Time to seroconversion during treatment | Baseline to Year 3
  The time to seroconversion in relation to exposure to study drug will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Inc., Foster City, California, United States

IPD SHARING:
Plan to Share IPD: No